CLINICAL TRIAL: NCT03652012
Title: Probing Cortical Excitability and Cognitive Function in Mild Cognitive Impairment With Transcranial Magnetic Stimulation
Brief Title: Probing Cortical Excitability and Cognitive Function With TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ying-hui Chou, Assistant Professor of Psychology, Cognition and Neural Systems Program, University of Arizona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1707654427
Record Dates: First submitted 2018-04-27; First posted 2018-08-29 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Dysfunction
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Mild Cognitive Impairment (Experimental): The following revised Mayo Clinic criteria for MCI (Petersen, et al. 2014) will be used: (1) cognitive concern expressed by a physician, informant, participant, or nurse; (2) impairment in 1 or more cognitive domains (memory, language, visuospatial skills, or executive functions); (3) essentially normal functional activities; and (4) absence of dementia. Individuals with MCI will have Mini-Mental State Exam (MMSE, Appendix 19) scores between 18 and 23 (inclusive) and have a Clinical Dementia Rating Scale score of 0.5.
  This group will undergo Transcranial Magnetic Stimulation (TMS) protocol.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Healthy Controls (Active Comparator): Participants who are matched for age and gender.
  This group will undergo Transcranial Magnetic Stimulation (TMS) protocol.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — TMS in a non-invasive brain stimulation technique. In this study, we will use TMS to excite brain tissue in the motor cortex and measure the subsequent motor response in the hand. This 'intervention' will be the same in both cohorts, as we are interested in how this motor response to TMS may vary across two distinct cohorts.

SUMMARY:
The overarching purpose of this study is to develop a technique that is capable of identifying neurophysiological biomarkers sensitive enough to detect preclinical dementia by integrating Transcranial Magnetic Stimulation (TMS) and Functional Magnetic Resonance Imaging (fMRI). More specifically, this project has two specific aims:

* 1. To characterize cortical excitability and its relation to cognitive function using single-pulse TMS paradigm in Mild Cognitive Impairment (MCI) and healthy older adults.
* 2. To delineate cortical plasticity and its association to cognitive function using repetitive TMS paradigm and resting-state fMRI in MCI and healthy older adults.

Techniques to artificially and precisely stimulate brain tissue are increasingly recognized as valuable tools both in clinical practice and in cognitive neuroscience studies among healthy individuals. Transcranial magnetic stimulation (TMS) is a non-invasive approach to stimulate the brain. Importantly, unlike other invasive brain stimulation techniques (e.g., surgical deep brain stimulation), no surgery, anesthesia, or sedation is involved. Instead, TMS involves placing a magnetic coil on the surface of the head. This coil then generates a magnetic field that is about the same strength as the magnetic field used by MRI machines, and when this magnetic field rapidly alternates, the neurons under the coil are excited.

Extensive guidelines have been published by experts in the field to ensure safe use, and the thousands of patients & research participants who have received TMS in compliance with these guidelines demonstrate the safety of this practice. Depending on the method of use, TMS is very versatile -- it can be used to study research questions pertaining to the neural circuitry of the brain, it can be used as a diagnostic device, and it can be used therapeutically to treat various neurological conditions.

In this study, the investigators intend to further study the potential for diagnostic applications of TMS. More specifically, TMS and brain imaging techniques will be used in combination in order to more sensitively diagnose dementia - perhaps even before symptoms emerge. Right now, there is no reliable method for doing so and it is difficult to distinguish between the forgetfulness of healthy aging and the early signs of disease. Our approach may provide a more sensitive diagnostic tool, which is likely to improve clinical outcomes.

DETAILED DESCRIPTION:
In total, 60 participants will be recruited to participate in this trial. The investigators aim to recruit 30 patients with MCI and 30 age-matched healthy adults. The age range for inclusion will be 18-80, and the mean age of the healthy cohort will be matched with the mean age of the MCI cohort. The following revised Mayo Clinic criteria for MCI will be used: (1) cognitive concern expressed by a physician, informant, participant, or nurse; (2) impairment in 1 or more cognitive domains (memory, language, visuospatial skills, or executive functions); (3) essentially normal functional activities; and (4) absence of dementia. Individuals with MCI will have Mini-Mental State Exam (MMSE, Appendix 19) scores between 18 and 23 (inclusive) and have a Clinical Dementia Rating Scale score of 0.5.

This study protocol comprises a single testing visit, comprised of four separate components: a) Resting-state fMRI, b) Single-pulse TMS paradigm, c) theta-burst rTMS paradigm, and d) a brief motor task performed on an iPad.

These tasks will be repeated before and after the theta-burst rTMS paradigm (c). Therefore, the testing visit is:

(a) --> (d) --> (b) --> (c) --> (b) --> (a) --> (d)

This protocol will enable investigators to study the following both before and after the rTMS paradigm: 1) connectivity patterns comprising the functional networks of the brain, 2) measures of cortical excitability derived from single-pulse TMS, and 3) upper extremity motor speed & acuity.

Transcranial Magnetic Stimulation:

Magnetic stimulation will be performed with a high-power MagPro X100 (MagVenture Inc. Denmark)(Appendix 11). When the TMS machine delivers stimuli, patients may feel and/or a clicking/tapping sensation under the coil. Participants will be given ear buds as an additional safety precaution to protect hearing during the TMS session. Prior to beginning the TMS session, the research team will make sure the participant is as comfortable as possible in the TMS chair.

Single Pulse TMS Paradigm:

First, the device will need to be calibrated for each individual because everybody has a different sensitivity to the magnetic fields generated by TMS. The TMS device will be calibrated to ensure the participant is receiving the lowest possible "dose". To do so, the TMS coil will be placed on the scalp directly above the region of the brain that is responsible for finger motions, which is a specific region of the motor cortex located on the pre-central gyrus. The TMS coil will then deliver pulses that incrementally escalate until a level is reached that causes their hand to twitch (specifically, thumb and pointer finger). This will be visually observed and recorded quantitatively with electromyography (EMG) sensors. The amount of energy required to make their hand twitch is called the "motor threshold" and it varies for everybody. This "motor threshold" will then be used to calibrate the machine for the TMS protocol.

A figure-of-eight TMS coil will be held over the motor cortex at the optimum scalp position to elicit motor-evoked potentials (MEPs) in the contralateral first dorsal interosseous (FDI) muscle. In addition to observing the finger movement visually, the investigators will also attach surface electromyography (EMG) electrodes to the skin on the right FDI. The electrodes will detect any activity in muscles, which will yield a more accurate measurement for personal "motor threshold". The exact location that elicits a motor response in the contralateral FDI is referred to as the "hot spot". This location will be recorded using the real-time TMS 3D Neuronavigation System (Localite TMS Navigator, Germany, http://www.localite.de/en/products/tms-navigator/#c572) to ensure testing consistency in the following trials. Localite is a software package used in conjunction with TMS equipment. It incorporates an infrared camera to record location of the TMS coil relative to the participants head. This allows researchers to reliably place coil in the same precise location throughout the session.

The resting motor threshold (RMT) is defined as the minimum stimulus intensity that produces a liminal MEP (about 50 μV in 50% of 10 trials) at rest. The active motor threshold (AMT) is generally defined as the minimum stimulus intensity that produces a liminal MEP (about 200 μV in 50% of 10 trials) during isometric contraction of the tested muscle. Both RMT and AMT will be expressed as a percentage of the magnetic stimulator maximal output. The RMT and AMT data from individual participants will serve as a baseline measure of excitability to guide the intensity of our following single-pulses and repetitive TMS protocols, respectively. This will be performed for the left hemisphere. The researchers will also use the Parameter Estimation Sequential Testing (PEST) algorithm to more efficiently identify the RMT and AMT.

After the motor threshold and "hot spot" is identified for the participant, the TMS coil will be placed over the "hot spot" that was previously recorded by the Localite Navigator software and set the stimulus intensity at 80% of the participants uniquely identified AMT. For example, if the active motor threshold of a specific individual is determined to be 40% of the MagPro's maximal output, then the device intensity will be set to 32% of maximal output for the single pulse protocol (32 equals 80% of 40%, the AMT in this example). At this time, 8 TMS pulses are applied (separated by 6 seconds) as the TMS coil is fixed on the "hot spot". This step is repeated in increasing increments (i.e., 10% of AMT) up to an intensity equivalent to 150% of the participant's AMT. This protocol consists of 64 single-pulse stimuli, which will be delivered repeatedly 6 seconds apart. This procedure is safe and follows standard single-pulses TMS protocols that have been published previously.

This single-pulses TMS protocol will be performed twice, both before and after the rTMS protocol. Each single-pulses TMS protocol will last approximately 30 minutes. Combined, this equates to 128 stimuli during the "Single Pulses TMS" paradigms. Throughout the single-pulse protocol, participants will be asked to touch their pinky and thumb fingers to provide a subtle background voluntary contraction. This will 'facilitate' the motor pathway and lower the threshold for stimulation intensity throughout the protocol.

rTMS:

In the repetitive TMS (rTMS) protocol, a patterned rTMS paradigm called intermittent theta burst stimulation (iTBS) will be used. The iTBS consists of three biphasic TMS stimuli presented at 50 Hz, repeated every 200 ms for 2 seconds at an intensity of 80% of AMT (e.g., if AMT is determined to be 40% of maximal output, TMS will be delivered at 32% for this protocol). Therefore, each stimulation train will last for two seconds (30 stimuli per train) with an inter-train interval of 8 s. This rTMS protocol is comprised of 10 iTBS trains, totaling 300 stimuli from the magnetic coil.

During this rTMS protocol, the coil will be placed over the "hotspot" of the left hemisphere. The rTMS protocol will only be performed once and it will last approximately 10 minutes.

MRI Protocols:

This will occur in the same building, in a room adjacent to the TMS device. For their safety, participants will be asked to leave all metal objects and personal items (e.g., wallet, phone, jewelry) in the waiting room of the MRI center before entering the scanner room. Participants will be asked to lie on their backs and remain still for the duration of the MRI scan. They will be given earplugs to dampen the noise and to protect their hearing while they are in the scanner. A Velcro strap may also be place over the forehead and foam pillows will be provided to minimize head movement during the scans. Every effort will be made to make participants as comfortable as possible during the scan, including blankets for warmth and cushions to be placed under the knees/back to reduce stress from lying on one's back.

Participants will be reminded prior to the scan that their participation is voluntary and they may signal to stop the scan at any time. There is an intercom system in the scanner, which will enable the participants to communicate with the MRI technician and member (s) of the research team for the entire duration that they are in the scanner. Additionally, they will be able to immediately stop the exam at any time, either by squeezing a signal ball placed in their hand, which will alert the MRI technician in the control room, or by raising their legs, which will be seen by the experimenter in the control room.

Importantly, no contrast agent will be used in our collection of MRI data. Also, all MRI data will be acquired in "resting-state" so participants will just be asked to relax and remain still for the duration of the scan.

More specifically, MRI data will be collected on a Siemens 3.0 Tesla Skyra Magnet equipped with a 32-channel head coil. Total scan time will be 30 minutes. The order of sequences will be as follows: localizer scan (62 seconds), a Structural MPRAGE (9 minutes), a resting-state fMRI scan (5 minutes), and a diffusion-tensor imaging (DTI) scan (14 minutes). The localizer will be collected using the following parameters - direction: inferior to superior, TR= 8.6 ms, echo time (TE)=4.0 ms, flip angle = 20, FOV=250 mm, 5 slices, 7 mm slice thickness. High-resolution structural images will be acquired using a T1-weighted spoiled gradient recalled (SPGR) sequence (TR= 22ms; TE= 5.4ms; FOV= 25.6cm; flip angle= 20°; in-plane matrix size= 256 x 256; slice thickness= 1mm; number of slices= 172). Whole-brain resting-state fMRI data will be collected using T2*-weighted echo-planar imaging (EPI) (TR= 1.5s; TE= 30ms; FOV= 25.6cm; flip angle= 90°; in-plane matrix size= 64 x 64; slice thickness= 4mm), resulting in functional data from 39 axial slices with isotropic voxels of 4mm3. During the resting-state fMRI scan, participants will fixate on a cross-hair with eyes open. DTI images will be acquired in the axial plane using a diffusion sensitized parallel EPI sequence that measures diffusion in 86 directions (b-factor= 1000 s/mm2; TR= 7s; TE= 82.5ms; field of view (FOV)= 25.6cm, matrix= 128 x 128, 2mm interleaved slices; parallel acceleration factor= 2).

The resting-state fMRI data will be preprocessed using a pipeline (http://wiki.biac.duke.edu/biac:analysis:resting_pipeline) and tools in the Oxford Centre for Functional MRI of the Brain Software Library (FSL version 5.0.5, www.fmrib.ox.ac.uk/fsl). The preprocessing steps include slice-time correction, MCFLIRT for motion correction, Brain Extraction Tool (BET) for brain extraction, and FLIRT for normalization to the MNI 152 T1 template (Montreal Neurological Institute, Montreal, Canada). The investigators will regress out signal from white matter and cerebrospinal fluid on the basis of masks created in FSL FAST and smoothed the data with a 5 mm kernel using FSL SUSAN. Temporal band-pass filtering will limit the data to frequencies in the 0.001 to 0.08 Hz band. Following the recommendation of Power et al., the investigators will perform motion scrubbing using a frame-wise displacement threshold of 0.5 and timecourse variance threshold (DVARS) of 0.5%

Behavioral Measure: Motor Task

The researchers will use iPads equipped with the digital computer software Cantab (Cambridge Cognition Ltd., England) for our behavioral measures. Cantab is a cloud-based, computerized cognitive assessment software that is a well-validated tool for academic research. The investigators intend to use 1) Motor Screening Task, 2) Paired Associates Learning Test (on a tablet) to measure functions of motor and memory, respectively.

Motor Screening Task requires the participants to touch the flashing cross, which is shown in different locations on the screen. The outcome measures include the accuracy of pointing and reaction time.

ELIGIBILITY:
Inclusion Criteria:

* The following revised Mayo Clinic criteria for MCI will be used: (1) cognitive concern expressed by a physician, informant, participant, or nurse; (2) impairment in 1 or more cognitive domains (memory, language, visuospatial skills, or executive functions); (3) essentially normal functional activities; and (4) absence of dementia. Individuals with MCI will have Mini-Mental State Exam (MMSE, Appendix 19) scores between 18 and 23 (inclusive) and have a Clinical Dementia Rating Scale score of 0.5.
* Health controls will be screened with MMSE

Exclusion Criteria:

* Contraindications to MRI
* Contraindications to TMS
* history of stroke
* clinical diagnosis of dementia
* diagnosis of neuropsychiatric disorder
* left handed

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sundman MH, Lim K, Ton That V, Mizell JM, Ugonna C, Rodriguez R, Chen NK, Fuglevand AJ, Liu Y, Wilson RC, Fellous JM, Rapcsak S, Chou YH. Transcranial magnetic stimulation reveals diminished homoeostatic metaplasticity in cognitively impaired adults. Brain Commun. 2020 Nov 27;2(2):fcaa203. doi: 10.1093/braincomms/fcaa203. eCollection 2020. PMID 33376989

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Cognitive Impairment: The following revised Mayo Clinic criteria for MCI (Petersen, et al. 2014) will be used: (1) cognitive concern expressed by a physician, informant, participant, or nurse; (2) impairment in 1 or more cognitive domains (memory, language, visuospatial skills, or executive functions); (3) essentially normal functional activities; and (4) absence of dementia. Individuals with MCI will have Mini-Mental State Exam (MMSE, Appendix 19) scores between 18 and 23 (inclusive) and have a Clinical Dementia Rating Scale score of 0.5.
  This group will undergo Transcranial Magnetic Stimulation (TMS) protocol.
  Transcranial Magnetic Stimulation (TMS): TMS in a non-invasive brain stimulation technique. In this study, we will use TMS to excite brain tissue in the motor cortex and measure the subsequent motor response in the hand. This 'intervention' will be the same in both cohorts, as we are interested in how this motor response to TMS may vary across two distinct cohorts.
- Healthy Controls: Participants who are matched for age and gender.
  This group will undergo Transcranial Magnetic Stimulation (TMS) protocol.
  Transcranial Magnetic Stimulation (TMS): TMS in a non-invasive brain stimulation technique. In this study, we will use TMS to excite brain tissue in the motor cortex and measure the subsequent motor response in the hand. This 'intervention' will be the same in both cohorts, as we are interested in how this motor response to TMS may vary across two distinct cohorts.
Period: Overall Study
Arm/Group | Mild Cognitive Impairment | Healthy Controls
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Cognitive Impairment | Healthy Controls | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (2.5) | 68.4 (3.2) | 69.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cortical Excitability: Resting Motor Threshold (RMT).
Description: Resting motor threshold (rMT) was determined using the Parameter Estimation by Sequential Testing (PEST) algorithm during a single-pulse transcranial magnetic stimulation (TMS) protocol. Surface electromyography (EMG) was used to record motor evoked potentials (MEPs) from the target muscle. rMT was defined as the minimum stimulation intensity over the motor cortex hotspot required to elicit an MEP of at least 50 μV in peak-to-peak amplitude in 50% of trials.
  Stimulation intensity on the TMS device is expressed as a percentage of the maximum stimulator output (MSO), which ranges from 1-100% on the TMS device. Accordingly, rMT values are also reported in %MSO.
Time Frame: Up to 10 minutes. This is a single day trial. Testing session will last a total of 3 hours.
Measure: Mean (Standard Deviation); unit: % of Max Stimulation Output (MSO)
Arm/Group | Mild Cognitive Impairment | Healthy Controls
Number analyzed (Participants) | 20 | 20
% of Max Stimulation Output (MSO) | 51.1 (6.6) | 51.8 (8.3)

2. Secondary Outcome: Cortical Excitability: Stimulus Response Curve. Measured With EMG, This Measures Motor Response to Various Intensities of Magnetic Pulse Stimuli
Description: Measured with surface EMG during single-pulse TMS paradigm. The outcome measure is derived from the varying Motor-Evoked Response potentials that are induced by variable TMS stimulation intensities. Specifically, this outcome measure is the slope of the stimulus-response curve, which is fitted to model the rise in MEP amplitude with rising TMS intensity.
Time Frame: Up to 30 minutes. This is a single day trial. Testing session will last a total of 3 hours.
Measure: Mean (Standard Error); unit: Slope
Groups:
- Mild Cognitive Impairment -- Active Muscle Condition: The following revised Mayo Clinic criteria for MCI (Petersen, et al. 2014) will be used: (1) cognitive concern expressed by a physician, informant, participant, or nurse; (2) impairment in 1 or more cognitive domains (memory, language, visuospatial skills, or executive functions); (3) essentially normal functional activities; and (4) absence of dementia. Individuals with MCI will have Mini-Mental State Exam (MMSE, Appendix 19) scores between 18 and 23 (inclusive) and have a Clinical Dementia Rating Scale score of 0.5.
  This group will undergo Transcranial Magnetic Stimulation (TMS) protocol.
  Transcranial Magnetic Stimulation (TMS): TMS in a non-invasive brain stimulation technique. In this study, we will use TMS to excite brain tissue in the motor cortex and measure the subsequent motor response in the hand. This 'intervention' will be the same in both cohorts, as we are interested in how this motor response to TMS may vary across two distinct cohorts. The motor response caused by the TMS pulse is referred to as the Motor Evoked Potential (MEP), which is measured from intrinsic hand muscles.
  This group provided a tonic voluntary muscle contraction (20% of their max force) in the target muscle during MEP acquisitions. We assessed MEP amplitude across different TMS intensities to model a stimulus-response curve.
- Healthy Controls -- Active Muscle Condition: Participants who are matched for age and gender.
  This group will undergo Transcranial Magnetic Stimulation (TMS) protocol.
  Transcranial Magnetic Stimulation (TMS): TMS in a non-invasive brain stimulation technique. In this study, we will use TMS to excite brain tissue in the motor cortex and measure the subsequent motor response in the hand. This 'intervention' will be the same in both cohorts, as we are interested in how this motor response to TMS may vary across two distinct cohorts. The motor response caused by the TMS pulse is referred to as the Motor Evoked Potential (MEP), which is measured from intrinsic hand muscles.
  This group provided a tonic voluntary muscle contraction (20% of their max force) in the target muscle during MEP acquisitions. We assessed MEP amplitude across different TMS intensities to model a stimulus-response curve.
- Mild Cognitive Impairment -- Rest Muscle Condition: The following revised Mayo Clinic criteria for MCI (Petersen, et al. 2014) will be used: (1) cognitive concern expressed by a physician, informant, participant, or nurse; (2) impairment in 1 or more cognitive domains (memory, language, visuospatial skills, or executive functions); (3) essentially normal functional activities; and (4) absence of dementia. Individuals with MCI will have Mini-Mental State Exam (MMSE, Appendix 19) scores between 18 and 23 (inclusive) and have a Clinical Dementia Rating Scale score of 0.5.
  This group will undergo Transcranial Magnetic Stimulation (TMS) protocol.
  Transcranial Magnetic Stimulation (TMS): TMS in a non-invasive brain stimulation technique. In this study, we will use TMS to excite brain tissue in the motor cortex and measure the subsequent motor response in the hand. This 'intervention' will be the same in both cohorts, as we are interested in how this motor response to TMS may vary across two distinct cohorts. The motor response caused by the TMS pulse is referred to as the Motor Evoked Potential (MEP), which is measured from intrinsic hand muscles.
  In this group, MEPs were acquired while the target muscle was at rest. We assessed MEP amplitude across different TMS intensities to model a stimulus-response curve.
- Healthy Controls -- Rest Muscle Condition: Participants who are matched for age and gender.
  This group will undergo Transcranial Magnetic Stimulation (TMS) protocol.
  Transcranial Magnetic Stimulation (TMS): TMS in a non-invasive brain stimulation technique. In this study, we will use TMS to excite brain tissue in the motor cortex and measure the subsequent motor response in the hand. This 'intervention' will be the same in both cohorts, as we are interested in how this motor response to TMS may vary across two distinct cohorts. The motor response caused by the TMS pulse is referred to as the Motor Evoked Potential (MEP), which is measured from intrinsic hand muscles.
  In this group, MEPs were acquired while the target muscle was at rest. We assessed MEP amplitude across different TMS intensities to model a stimulus-response curve.
Arm/Group | Mild Cognitive Impairment -- Active Muscle Condition | Healthy Controls -- Active Muscle Condition | Mild Cognitive Impairment -- Rest Muscle Condition | Healthy Controls -- Rest Muscle Condition
Number analyzed (Participants) | 10 | 10 | 10 | 10
Slope | 56.04 (7.14) | 122.04 (27.93) | 65.05 (14.41) | 107.45 (40.99)
Statistical Analysis 1: Comparison: Mild Cognitive Impairment -- Active Muscle Condition vs Healthy Controls -- Active Muscle Condition vs Mild Cognitive Impairment -- Rest Muscle Condition vs Healthy Controls -- Rest Muscle Condition; We conducted a two-way factorial ANOVA (Group x Condition). "Group" has two levels: MCI and Healthy controls. "Condition" has two levels: active muscle contraction and rest. As multiple parameters were assessed from the stimulus-response curve, a Bonferroni-adjusted alpha threshold of α = 0.0125 was applied to account for multiple comparisons when assessing this outcome measure; Test type: Superiority; p = 0.044, ANOVA — As multiple parameters were assessed from the stimulus-response curve, a Bonferroni-adjusted alpha threshold of α = 0.0125 was applied to account for multiple comparisons when assessing this outcome measure; Mean Difference (Final Values) = 54.2, 95% CI 2-sided [1.54 to 106.85] — Mean difference (Healthy Controls - MCI)
Statistical Analysis 2: Comparison: Mild Cognitive Impairment -- Active Muscle Condition vs Healthy Controls -- Active Muscle Condition vs Mild Cognitive Impairment -- Rest Muscle Condition vs Healthy Controls -- Rest Muscle Condition; We conducted a two-way factorial ANOVA (Group x Condition). "Group" has two levels: MCI and Healthy controls. "Condition" has two levels: active muscle contraction and rest. As multiple parameters were assessed from the stimulus-response curve, a Bonferroni-adjusted alpha threshold of α = 0.0125 was applied to account for multiple comparisons when assessing this outcome measure. The results presented here reflect the main effect of Condition on the slope of the stimulus-response curve; Test type: Superiority; p = 0.912, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-51.87 to 57.47] — Mean difference in slope of the stimulus-response curve by muscle contraction condition (Active - Rest)

3. Secondary Outcome: Cortical Excitability: Cortical Silent Period. Measured With EMG, This is a Direct Measure of Cortical Inhibition.
Description: Measured with surface EMG during single-pulse TMS paradigm. Participants will be asked to voluntary contract hand muscle, at 20% of their maximum contraction force. A TMS pulse is applied while participants are applying this voluntary contraction. The cortical silent period is defined as the duration between the observed motor evoked potential and the resumption of muscle voluntary contraction.
Time Frame: Up to 10 minutes. This is a single day trial. Testing session will last a total of 3 hours.
Measure: Mean (Standard Error); unit: Duration (milliseconds)
Arm/Group | Mild Cognitive Impairment | Healthy Controls
Number analyzed (Participants) | 20 | 20
Duration (milliseconds) | 131.30 (10.24) | 151.91 (6.73)
Statistical Analysis 1: Comparison: Mild Cognitive Impairment vs Healthy Controls; Test type: Superiority; p = 0.1021, t-test, 2 sided; No adjustment for multiple comparisons; Mean Difference (Final Values) = 20.6, 95% CI 2-sided [-4.33 to 45.54] — Mean cortical silent period (CSP; units = milliseconds) in the CN group minus mean CSP in the MCI group. Positive values indicate a longer cortical silent period in the control group

4. Secondary Outcome: Baseline Functional Magnetic Resonance Imaging (fMRI) to Observe Functional Activation of Brain Networks Prior to Intervention.
Description: This resting state fMRI scan measured functional connectivity patterns at baseline prior to a non-invasive brain stimulation protocol targeting the primary motor cortex (M1). We measured resting-state functional connectivity between the left M1 and the left somatosensory cortex (S1). Functional connectivity was quantified using Pearson correlation coefficients between the time series of the two regions, which were then Fisher Z-transformed to normalize the distribution. The unit of measure is the Fisher Z-transformed correlation value (unitless).
Time Frame: Up to 30 minutes. This is a single day trial. Testing session will last a total of 3 hours.
Measure: Mean (Standard Deviation); unit: Fisher Z correlation (unitless)
Groups:
- Mild Cognitive Impairment: The following revised Mayo Clinic criteria for MCI (Petersen, et al. 2014) will be used: (1) cognitive concern expressed by a physician, informant, participant, or nurse; (2) impairment in 1 or more cognitive domains (memory, language, visuospatial skills, or executive functions); (3) essentially normal functional activities; and (4) absence of dementia. Individuals with MCI will have Mini-Mental State Exam (MMSE, Appendix 19) scores between 18 and 23 (inclusive) and have a Clinical Dementia Rating Scale score of 0.5.
- Healthy Controls: Cognitive normal participants who are matched for age and gender.
Arm/Group | Mild Cognitive Impairment | Healthy Controls
Number analyzed (Participants) | 10 | 10
Fisher Z correlation (unitless) | 0.741 (0.314) | 0.534 (0.282)
Statistical Analysis 1: Comparison: Mild Cognitive Impairment vs Healthy Controls; Test type: Superiority; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = .208, 95% CI 2-sided [-0.113 to 0.529]

5. Secondary Outcome: Post Functional Magnetic Resonance Imaging (fMRI): Change in Functional Connectivity Following TMS.
Description: This outcome measure assesses the change in resting-state functional connectivity between the left primary motor cortex (M1) and the left somatosensory cortex (S1), measured immediately after TMS was applied to the left M1. Functional connectivity was quantified using Pearson correlation coefficients between the time series of the two regions, which were then Fisher Z-transformed to normalize the distribution. The unit of measure is the Fisher Z-transformed correlation value (unitless). Positive values reflect an increase in functional connectivity from baseline, whereas negative values indicate a decrease.
Time Frame: Up to 30 minutes. This is a single day trial. Testing session will last a total of 3 hours.
Measure: Mean (Standard Deviation); unit: Fisher Z correlation (unitless)
Arm/Group | Mild Cognitive Impairment | Healthy Controls
Number analyzed (Participants) | 10 | 10
Fisher Z correlation (unitless) | -0.068 (0.302) | -0.060 (0.526)
Statistical Analysis 1: Comparison: Mild Cognitive Impairment vs Healthy Controls; Test type: Superiority; p = 0.97, t-test, 2 sided; Mean Difference (Net) = 0.0078, 95% CI 2-sided [-0.51 to 0.50]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Mild Cognitive Impairment | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT03652012/Prot_SAP_001.pdf